CLINICAL TRIAL: NCT02434497
Title: An Open-Label Long-Term Extension to the Randomized, Double-blind, Placebo-controlled, Multi-center, Cross-over Study of Rosuvastatin in Children and Adolescents (Aged 6 to <18 Years) With Homozygous Familial Hypercholesterolemia (HoFH)
Brief Title: A Study to Evaluate the Safety of Rosuvastatin in Children and Adolescents With Homozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D356NC00001
Record Dates: First submitted 2015-04-07; First posted 2015-05-05 (Estimated); Results first posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Homozygous Familial Hypercholesterolemia (HoFH)
Keywords: LDL-C; HoFH; Hyperlipidemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Hyperlipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): One treatment period for all patients (<1 year and 10 months), with the possibility to up-titrate dose to 40 mg of rosuvastatin for non-Asian patients.
  Interventions: Drug: Rosuvastatin 20mg

INTERVENTIONS:
Drug: Rosuvastatin 20mg — Active drug 1 or 2 tablets will be taken taken orally, QD, either in the morning or in the evening

SUMMARY:
The purpose of the study is to evaluate the safety of Rosuvastatin in Children and Adolescents with Homozygous Familial Hypercholesterolemia.

DETAILED DESCRIPTION:
This is a long-term extension (LTE) to the randomized, double-blind, cross-over study of rosuvastatin 20 mg once daily (QD) versus placebo QD in children and adolescents (aged from 6 to <18 years) with homozygous familial hypercholesterolemia (HoFH) (Study D3561C00004).

The study is designed to assess the long-term safety and tolerability of rosuvastatin 20 mg in pediatric patients with HoFH.

In this study all patients will receive rosuvastatin 20 mg QD. Investigators will also be permitted to titrate the dose of rosuvastatin from 20 to 40 mg per day if they feel it is warranted to more aggressively treat patients' elevated LDL-C levels. This up-titration will not be permitted in Asian patients. Pharmacokinetic data of the trough plasma exposure of rosuvastatin will also be assessed for the pediatric patients with HoFH taking a daily dose of rosuvastatin 40 mg.

The primary outcome measures to be assessed include 1) Adverse events, including:

* The frequency and severity of adverse events,
* Rate of discontinuations due to adverse events,
* Abnormal serum and urine laboratory values, electrocardiograms (ECGs), physical examinations, and vital signs; and 2) Assessments of growth.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to any study related procedures being performed, provision of written informed consent from a parent/both parents or guardian and statement of assent from the child or adolescent (if required by Institutional Review Board [IRB] or Independent Ethics Committee [IEC] according to local regulations and guidelines). Study D3561C00004 participants who have had their 18th birthday (adults) will be required to provide written informed consent. Communication should take place between the Investigator, patient/guardian and child/adolescent to confirm understanding and required compliance with the requirements of the study.
2. Male and female children and adolescents who were aged 6 to <18 years at the onset of Study D3561C00004 (even if they had their 18th birthday during that study) with:

   * Documentation of genetic testing confirming 2 mutated alleles of the LDL receptor gene locus; and/or
   * Documented untreated LDL C >500 mg/dL (12.9 mmol/L) and TG <400 mg/dL (4.5 mmol/L) and at least 1 of the following criteria:

     * Tendinous and/or cutaneous xanthoma prior to 10 years of age; or
     * Documentation of HeFH in both parents by:
   * genetic and/or
   * clinical criteria
3. Negative pregnancy test (b human chorionic gonadotropin analysis) prior to baseline in females of child bearing potential:

   * Female patients of child bearing potential must adhere to a pregnancy prevention method (abstinence, chemical, or mechanical) during the study and 3 months following the last dose;
   * Male patients should refrain from fathering a child (including sperm donation) during the study and up to 3 months following the last dose; and
4. Were taking study drug at the end of Study D3561C00004 and are willing to follow all study procedures including adherence to dietary guidelines, study visits, fasting blood draws, and compliance with study treatment regimens.

Exclusion Criteria:

1. History of statin inducted myopathy or serious hypersensitivity reaction to other HMG CoA reductase inhibitors (statins), including rosuvastatin, at Visit 1 of Study D3561C00004.
2. Fasting serum glucose of >9.99 mmol/L (180 mg/dL) or glycosylated hemoglobin >9% during Study D3561C00004 or patients with a history of diabetic ketoacidosis within the past year.
3. Uncontrolled hypothyroidism defined as thyroid stimulating hormone >1.5 times the upper limit of normal (ULN) at any time during Study D3561C00004.
4. Evidence of active liver disease or hepatic dysfunction (except a confirmed diagnosis of Gilbert's disease) as defined as non-transient elevations of ALT or AST elevations ≥3 times the ULN or non-transient total bilirubin ≥2 times the ULN during the Study D3561C00004.
5. Definite or suspected personal history or family history of clinically significant adverse drug reactions (ADRs), or hypersensitivity to drugs with a similar chemical structure to rosuvastatin as well as other statins.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2015-06-06 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2016-11-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Research Site, Brussels (Woluwé-St-Lambert), Belgium
- Research Site, Chicoutimi, Quebec, Canada
- Research Site, Copenhagen, Denmark
- Research Site, Halfa, Israel
- Research Site, Kubang Kerian, Malaysia
- Research Site, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The nine (9) patients recruited were all participants in the D3561C00004 HYDRA study (NCT02226198) four came from Sequence A and five from Sequence B
Groups:
- Overall: All patients
Period: Overall Study
Arm/Group | Overall
Started | 9
Completed | 4
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Overall
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (2.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Experianced Adverse Events and Serious Adverse Events
Time Frame: 96 weeks
Measure: Number; unit: participants
Groups:
- Full Analysis Set: Full analysis set, comprised of patient who received at least one dose of study drug.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
participants | 5

2. Primary Outcome: Safety and Tolerability in Terms of Number of Participants Who Had Adverse Events, Discontinuations Due to Adverse Events
Time Frame: 96 weeks
Measure: Number; unit: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
participants | 0

3. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Basophils/Leukocytes (%) >Upper Limite of Normal (ULN)
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Groups:
- Sequence A: Rosuva/Placebo in the D3561C00004 cross-over phase
- Sequence B: Placebo/Rosuva in the D3561C00004 cross-over phase
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 1 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

4. Primary Outcome: Safety and Tolerability in Terms of Growth, Height
Time Frame: 96 weeks
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
cm
  Baseline | 142.5 (23.57) | 136.8 (15.02)
  Week 6 | 143.5 (23.57) | 136.8 (15.32)
  Week 12 | 144.0 (23.90) | 137.6 (14.94)
  Week 18 | 145.3 (23.56) | 138.0 (14.83)
  Week 24 | 145.8 (24.02) | 139.2 (15.74)
  Week 36 | 147.0 (24.15) | 140.6 (15.61)
  Week 48 | 148.8 (24.25) | 142.2 (15.21)
  Week 60 | 158.0 (19.47) | 144.0 (16.37)
  Week 72 | 159.0 (20.22) | 145.0 (15.12)
  Week 84 | 159.7 (20.43) | 148.3 (17.27)
  Week 96 | 165.0 (25.46) | 138.0 (12.73)

5. Primary Outcome: Safety and Tolerability in Terms of Abnormalitites in Sexual Maturation
Time Frame: 96 weeks
Measure: Number; unit: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
participants | 0

6. Primary Outcome: Safety and Tolerability in Terms of Growth, Height SD-score (or Z-score)
Description: Height z-score is a dimensionless quantity derived by subtracting the population mean from the individual raw score, and then deviding the difference by the pouulation SD of the reference population. This indicates how many SDs and observation is above or below the general population mean.
Time Frame: 96 weeks
Measure: Mean (Standard Deviation); unit: standard deviations
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
standard deviations
  Baseline | -0.43 (2.025) | -1.05 (1.787)
  Week 6 | -0.48 (1.911) | -1.05 (1.871)
  Week 12 | -0.41 (1.975) | -1.19 (1.709)
  Week 18 | -0.43 (1.610) | -1.14 (1.705)
  Week 24 | -0.60 (1.730) | -0.96 (1.670)
  Week 36 | -0.43 (1.836) | -0.76 (1.727)
  Week 48 | -0.16 (1.781) | -0.72 (1.729)
  Week 60 | 0.05 (1.757) | -1.04 (1.604)
  Week 72 | 0.00 (1.635) | -0.87 (1.604)
  Week 84 | 0.08 (1.734) | -0.33 (1.627)
  Week 96 | 1.18 (0.436) | -0.51 (0.886)

7. Primary Outcome: Safety and Tolerability in Terms of Growth, Weight
Time Frame: 96 weeks
Measure: Mean (Standard Deviation); unit: kg
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
kg
  Baseline | 36.25 (14.719) | 37.42 (16.089)
  Week 6 | 37.20 (16.230) | 38.02 (16.700)
  Week 12 | 37.93 (17.110) | 38.16 (17.501)
  Week 18 | 38.85 (17.633) | 38.40 (16.688)
  Week 24 | 39.15 (17.521) | 39.00 (16.704)
  Week 36 | 39.98 (18.293) | 39.88 (15.015)
  Week 48 | 41.00 (17.579) | 41.16 (16.045)
  Week 60 | 48.47 (16.933) | 41.80 (15.656)
  Week 72 | 48.43 (16.393) | 42.10 (17.047)
  Week 84 | 50.17 (16.737) | 45.28 (19.143)
  Week 96 | 57.35 (16.476) | 33.55 (2.192)

8. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Alanine Aminotransferase (U/L) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 1 (14.94)
  Week 18 | 0 (23.56) | 1 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 1 (15.61)
  Week 48 | 0 (24.25) | 1 (15.21)
  Week 60 | 0 (19.47) | 1 (16.37)
  Week 72 | 0 (20.22) | 1 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

9. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Albumin (g/dL) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 1 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 1 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

10. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Aspartate Aminotransferase (U/L) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 1 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

11. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Bicarbonate (Mol/L) <LLN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 1 (15.32)
  Week 12 | 1 (23.90) | 1 (14.94)
  Week 18 | 0 (23.56) | 1 (14.83)
  Week 24 | 1 (24.02) | 1 (15.74)
  Week 36 | 1 (24.15) | 2 (15.61)
  Week 48 | 1 (24.25) | 1 (15.21)
  Week 60 | 1 (19.47) | 3 (16.37)
  Week 72 | 2 (20.22) | 1 (15.12)
  Week 84 | 1 (20.43) | 1 (17.27)
  Week 96 | 0 (25.46) | 1 (12.73)

12. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Bicarbonate (Mol/L) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 1 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

13. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Ery. Mean Corpuscular HGB Concentration (g/dL) <LLN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 2 (23.57) | 3 (15.02)
  Week 6 | 0 (23.57) | 2 (15.32)
  Week 12 | 2 (23.90) | 2 (14.94)
  Week 18 | 1 (23.56) | 2 (14.83)
  Week 24 | 2 (24.02) | 3 (15.74)
  Week 36 | 1 (24.15) | 3 (15.61)
  Week 48 | 1 (24.25) | 4 (15.21)
  Week 60 | 1 (19.47) | 4 (16.37)
  Week 72 | 2 (20.22) | 3 (15.12)
  Week 84 | 2 (20.43) | 3 (17.27)
  Week 96 | 0 (25.46) | 1 (12.73)

14. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Ery. Mean Corpuscular HGB (pg) <LLN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 1 (23.57) | 3 (15.02)
  Week 6 | 1 (23.57) | 2 (15.32)
  Week 12 | 1 (23.90) | 2 (14.94)
  Week 18 | 1 (23.56) | 2 (14.83)
  Week 24 | 1 (24.02) | 2 (15.74)
  Week 36 | 1 (24.15) | 2 (15.61)
  Week 48 | 1 (24.25) | 3 (15.21)
  Week 60 | 0 (19.47) | 3 (16.37)
  Week 72 | 0 (20.22) | 3 (15.12)
  Week 84 | 0 (20.43) | 3 (17.27)
  Week 96 | 2 (25.46) | 1 (12.73)

15. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Ery. Mean Corpuscular Volume (fL) <LLN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 1 (23.57) | 2 (15.02)
  Week 6 | 1 (23.57) | 2 (15.32)
  Week 12 | 1 (23.90) | 2 (14.94)
  Week 18 | 1 (23.56) | 2 (14.83)
  Week 24 | 1 (24.02) | 2 (15.74)
  Week 36 | 1 (24.15) | 2 (15.61)
  Week 48 | 1 (24.25) | 2 (15.21)
  Week 60 | 0 (19.47) | 2 (16.37)
  Week 72 | 0 (20.22) | 3 (15.12)
  Week 84 | 0 (20.43) | 3 (17.27)
  Week 96 | 2 (25.46) | 1 (12.73)

16. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Ery. Mean Corpuscular Volume (fL) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 1 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

17. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Erythrocytes (10^12/L) <LLN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 1 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 1 (14.94)
  Week 18 | 0 (23.56) | 1 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 1 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 1 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

18. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Erythrocytes (10^12/L) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 1 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 1 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 1 (24.02) | 2 (15.74)
  Week 36 | 0 (24.15) | 2 (15.61)
  Week 48 | 0 (24.25) | 1 (15.21)
  Week 60 | 0 (19.47) | 1 (16.37)
  Week 72 | 0 (20.22) | 2 (15.12)
  Week 84 | 0 (20.43) | 1 (17.27)
  Week 96 | 0 (25.46) | 1 (12.73)

19. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Hematocrit (%) <LLN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 2 (23.57) | 2 (15.02)
  Week 6 | 2 (23.57) | 3 (15.32)
  Week 12 | 1 (23.90) | 2 (14.94)
  Week 18 | 1 (23.56) | 3 (14.83)
  Week 24 | 0 (24.02) | 1 (15.74)
  Week 36 | 1 (24.15) | 1 (15.61)
  Week 48 | 0 (24.25) | 2 (15.21)
  Week 60 | 0 (19.47) | 2 (16.37)
  Week 72 | 0 (20.22) | 1 (15.12)
  Week 84 | 0 (20.43) | 1 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

20. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Hemoglobin (g/dL) <LLN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 2 (23.57) | 3 (15.02)
  Week 6 | 2 (23.57) | 3 (15.32)
  Week 12 | 1 (23.90) | 3 (14.94)
  Week 18 | 1 (23.56) | 3 (14.83)
  Week 24 | 0 (24.02) | 2 (15.74)
  Week 36 | 1 (24.15) | 3 (15.61)
  Week 48 | 1 (24.25) | 3 (15.21)
  Week 60 | 0 (19.47) | 3 (16.37)
  Week 72 | 0 (20.22) | 3 (15.12)
  Week 84 | 0 (20.43) | 3 (17.27)
  Week 96 | 0 (25.46) | 1 (12.73)

21. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Leukocytes >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 1 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

22. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Lymphocytes/Leukocytes (%) <LLN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 1 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

23. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Lymphocytes/Leukocytes (%) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 1 (15.02)
  Week 6 | 0 (23.57) | 1 (15.32)
  Week 12 | 0 (23.90) | 1 (14.94)
  Week 18 | 0 (23.56) | 1 (14.83)
  Week 24 | 0 (24.02) | 1 (15.74)
  Week 36 | 0 (24.15) | 1 (15.61)
  Week 48 | 0 (24.25) | 1 (15.21)
  Week 60 | 0 (19.47) | 1 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

24. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Monocytes/Leukocytes (%) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 1 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

25. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Platelets (10^9/L) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 1 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 1 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 1 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 1 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

26. Secondary Outcome: Percent Change in LDL-C From End of Placebo of D3561C00004 to the End of D356NC00001, Repeated Measures Analysis
Time Frame: Up to 22 months
Measure: Geometric Mean (95% Confidence Interval); unit: % change from baseline LDL-C
Units Other Than Participants: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
% change from baseline LDL-C
  Visit 1 | -21.0 [-32.1 to -8.0]
  Visit 2 | -18.6 [-28.4 to -7.4]
  Visit 3 | -14.7 [-25.2 to -2.8]
  Visit 4 | -12.1 [-23.8 to 1.4]
  Visit 5 | -21.3 [-33.7 to -6.6]
  Visit 6 | -20.5 [-33.6 to -4.8]
  Visit 7 | -12.4 [-28.2 to 7.0]

27. Secondary Outcome: Percent Change in HDL-C From End of Placebo of D3561C00004 to the End of D356NC00001, Repeated Measures Analysis
Time Frame: Up to 22 months
Measure: Geometric Mean (95% Confidence Interval); unit: % change from baseline HDL-C
Units Other Than Participants: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
% change from baseline HDL-C
  Visit 1 | 12.3 [1.3 to 24.5]
  Visit 2 | 19.0 [6.2 to 33.4]
  Visit 3 | 5.2 [-8.4 to 20.8]
  Visit 4 | 4.4 [-10.8 to 22.2]
  Visit 5 | 4.4 [-12.7 to 24.9]
  Visit 6 | 9.4 [-9.4 to 32.1]
  Visit 7 | 3.8 [-13.1 to 23.9]

28. Secondary Outcome: Percent Change in Total Cholesterol (TC) From End of Placebo of D3561C00004 to the End of D356NC00001, Repeated Measures Analysis
Time Frame: Up to 22 months
Measure: Geometric Mean (95% Confidence Interval); unit: % change from baseline TC
Units Other Than Participants: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
% change from baseline TC
  Visit 1 | -19.4 [-29.7 to -7.6]
  Visit 2 | -16.8 [-25.7 to -6.8]
  Visit 3 | -14.0 [-23.6 to -3.3]
  Visit 4 | -11.8 [-22.3 to 0.1]
  Visit 5 | -19.9 [-31.1 to -6.9]
  Visit 6 | -18.3 [-30.2 to -4.3]
  Visit 7 | -11.9 [-26.3 to 5.2]

29. Secondary Outcome: Percent Change in Triglycerides (TG) From End of Placebo of D3561C00004 to the End of D356NC00001, Repeated Measures Analysis
Time Frame: Up to 22 months
Measure: Geometric Mean (95% Confidence Interval); unit: % change from baseline TG
Units Other Than Participants: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
% change from baseline TG
  Visit 1 | -17.3 [-31.9 to 0.5]
  Visit 2 | -17.4 [-34.2 to 3.8]
  Visit 3 | -16.2 [-36.1 to 10.1]
  Visit 4 | -22.0 [-42.8 to 6.5]
  Visit 5 | -23.3 [-45.0 to 7.1]
  Visit 6 | -21.7 [-43.4 to 8.4]
  Visit 7 | -28.5 [-47.0 to -3.6]

30. Secondary Outcome: Percent Change in Non-HDL-C From End of Placebo of D3561C00004 to the End of D356NC00001, Repeated Measures Analysis
Time Frame: Up to 22 months
Measure: Geometric Mean (95% Confidence Interval); unit: % change from baseline Non-HDL-C
Units Other Than Participants: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
% change from baseline Non-HDL-C
  Visit 1 | -21.7 [-32.7 to -9.0]
  Visit 2 | -19.2 [-28.8 to -8.3]
  Visit 3 | -15.7 [-25.7 to -4.3]
  Visit 4 | -13.3 [-24.3 to -0.7]
  Visit 5 | -22.1 [-33.8 to -8.4]
  Visit 6 | -21.0 [-33.2 to -6.5]
  Visit 7 | -13.2 [-28.1 to 4.8]

31. Secondary Outcome: Percent Change in LDL-C/HDL-C From End of Placebo of D3561C00004 to the End of D356NC00001, Repeated Measures Analysis
Time Frame: Up to 22 months
Measure: Geometric Mean (95% Confidence Interval); unit: % change from baseline LDL-C/HDL-C
Units Other Than Participants: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
% change from baseline LDL-C/HDL-C
  Visit 1 | -39.4 [-51.6 to -24.1]
  Visit 2 | -41.2 [-52.8 to -26.9]
  Visit 3 | -36.1 [-48.8 to -20.2]
  Visit 4 | -35.0 [-49.5 to -16.4]
  Visit 5 | -48.6 [-61.3 to -31.7]
  Visit 6 | -42.2 [-57.2 to -21.9]
  Visit 7 | -27.8 [-47.4 to -0.9]

32. Secondary Outcome: Percent Change in TC/HDL-C From End of Placebo of D3561C00004 to the End of D356NC00001, Repeated Measures Analysis
Time Frame: Up to 22 months
Measure: Geometric Mean (95% Confidence Interval); unit: % change from baseline TC/HDL-C
Units Other Than Participants: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
% change from baseline TC/HDL-C
  Visit 1 | -30.6 [-38.3 to -21.9]
  Visit 2 | -29.4 [-38.5 to -18.9]
  Visit 3 | -20.5 [-32.0 to -7.0]
  Visit 4 | -16.6 [-30.7 to 0.4]
  Visit 5 | -24.1 [-38.6 to -6.2]
  Visit 6 | -29.2 [-43.2 to -11.7]
  Visit 7 | -15.6 [-33.7 to 7.5]

33. Secondary Outcome: Percent Change in Non-HDL-C/HDL-C From End of Placebo of D3561C00004 to the End of D356NC00001, Repeated Measures Analysis
Time Frame: Up to 22 months
Measure: Geometric Mean (95% Confidence Interval); unit: % change from baseline Non-HDL-C/HDL-C
Units Other Than Participants: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
% change from baseline Non-HDL-C/HDL-C
  Visit 1 | -32.9 [-41.2 to -23.3]
  Visit 2 | -31.5 [-41.2 to -20.3]
  Visit 3 | -22.3 [-34.3 to -8.1]
  Visit 4 | -18.1 [-32.8 to -0.3]
  Visit 5 | -26.3 [-41.3 to -7.4]
  Visit 6 | -31.8 [-46.0 to -13.9]
  Visit 7 | -17.6 [-36.2 to 6.5]

34. Secondary Outcome: Percent Change in ApoB From End of Placebo of D3561C00004 to the End of D356NC00001, Repeated Measures Analysis
Time Frame: Up to 22 months
Measure: Geometric Mean (95% Confidence Interval); unit: % change from baseline ApoB
Units Other Than Participants: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
% change from baseline ApoB
  Visit 1 | -20.5 [-29.8 to -9.9]
  Visit 2 | -18.7 [-26.7 to -9.8]
  Visit 3 | -15.2 [-23.9 to -5.6]
  Visit 4 | -10.5 [-20.4 to 0.5]
  Visit 5 | -17.2 [-27.9 to -4.9]
  Visit 6 | -19.2 [-30.2 to -6.5]
  Visit 7 | -9.5 [-23.5 to 7.2]

35. Secondary Outcome: Percent Change in ApoA-1 From End of Placebo of D3561C00004 to the End of D356NC00001, Repeated Measures Analysis
Time Frame: Up to 22 months
Measure: Geometric Mean (95% Confidence Interval); unit: % change from baseline ApoA-1
Units Other Than Participants: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
% change from baseline ApoA-1
  Visit 1 | 8.0 [0.0 to 16.6]
  Visit 2 | 7.0 [-2.3 to 17.1]
  Visit 3 | 5.3 [-4.9 to 16.7]
  Visit 4 | 6.5 [-5.3 to 19.7]
  Visit 5 | 1.0 [-11.5 to 15.3]
  Visit 6 | 10.7 [-2.6 to 25.7]
  Visit 7 | 1.6 [-12.9 to 18.4]

36. Secondary Outcome: Percent Change in ApoB/ApoA-1 From End of Placebo of D3561C00004 to the End of D356NC00001, Repeated Measures Analysis
Time Frame: Up to 22 months
Measure: Geometric Mean (95% Confidence Interval); unit: % change from baseline ApoB/ApoA-1
Units Other Than Participants: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 9
% change from baseline ApoB/ApoA-1
  Visit 1 | -23.3 [-34.3 to -10.5]
  Visit 2 | -22.1 [-32.7 to -9.8]
  Visit 3 | -18.9 [-31.2 to -4.4]
  Visit 4 | -15.7 [-30.2 to 1.7]
  Visit 5 | -17.0 [-33.1 to 2.8]
  Visit 6 | -26.0 [-41.1 to -7.0]
  Visit 7 | -14.7 [-33.7 to 9.7]

37. Secondary Outcome: Pharmacokinetic Profile in Terms of Trough Concentrations in Pediatric HoFH Taking a Daily Dose of Rosuvastatin 40mg
Time Frame: Up to 22 months
Measure: Number; unit: ng/mL
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 1
ng/mL
  Day 292 | 9.00
  Day 376 | 7.14

38. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Blood Urea Nitrogen (mg/dL) <LLN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 1 (23.57) | 0 (15.02)
  Week 6 | 1 (23.57) | 0 (15.32)
  Week 12 | 1 (23.90) | 0 (14.94)
  Week 18 | 1 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 1 (15.61)
  Week 48 | 1 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

39. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Chloride (mmol/L) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 1 (15.02)
  Week 6 | 0 (23.57) | 1 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 1 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 1 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 1 (16.37)
  Week 72 | 0 (20.22) | 1 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

40. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Creatine Kinase (U/L) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 1 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 1 (24.02) | 0 (15.74)
  Week 36 | 1 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 1 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 1 (25.46) | 0 (12.73)

41. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Glucose (mg/dL) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 1 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 1 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

42. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Lactate Dehydrogenase (U/L) <LLN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 1 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

43. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Phosphate (mg/dL) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 1 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 1 (15.12)
  Week 84 | 0 (20.43) | 1 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

44. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Protein (g/dL) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 1 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 1 (15.74)
  Week 36 | 1 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

45. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Sodium (mmol/L) <LLN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 2 (23.57) | 0 (15.02)
  Week 6 | 1 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 3 (23.56) | 1 (14.83)
  Week 24 | 0 (24.02) | 1 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 1 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 1 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

46. Primary Outcome: Safety and Tolerability in Terms of Abnormal Serum Laboratory Values, Urate (mg/dL) >ULN
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 1 (23.57) | 0 (15.02)
  Week 6 | 1 (23.57) | 1 (15.32)
  Week 12 | 1 (23.90) | 0 (14.94)
  Week 18 | 1 (23.56) | 1 (14.83)
  Week 24 | 1 (24.02) | 1 (15.74)
  Week 36 | 1 (24.15) | 1 (15.61)
  Week 48 | 1 (24.25) | 1 (15.21)
  Week 60 | 1 (19.47) | 1 (16.37)
  Week 72 | 1 (20.22) | 1 (15.12)
  Week 84 | 1 (20.43) | 1 (17.27)
  Week 96 | 1 (25.46) | 0 (12.73)

47. Primary Outcome: Safety and Tolerability in Terms of Abnormal Urine Laboratory Values, Urine Ketones
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 1 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 1 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 1 (25.46) | 0 (12.73)

48. Primary Outcome: Safety and Tolerability in Terms of Abnormal Urine Laboratory Values, Urine Occult Blood
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 1 (23.57) | 1 (15.02)
  Week 6 | 2 (23.57) | 1 (15.32)
  Week 12 | 1 (23.90) | 2 (14.94)
  Week 18 | 1 (23.56) | 1 (14.83)
  Week 24 | 1 (24.02) | 1 (15.74)
  Week 36 | 1 (24.15) | 1 (15.61)
  Week 48 | 1 (24.25) | 1 (15.21)
  Week 60 | 1 (19.47) | 1 (16.37)
  Week 72 | 2 (20.22) | 1 (15.12)
  Week 84 | 1 (20.43) | 1 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

49. Primary Outcome: Safety and Tolerability in Terms of Abnormal Urine Laboratory Values, Urine Protein
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 2 (23.57) | 1 (15.02)
  Week 6 | 1 (23.57) | 1 (15.32)
  Week 12 | 2 (23.90) | 1 (14.94)
  Week 18 | 1 (23.56) | 0 (14.83)
  Week 24 | 2 (24.02) | 1 (15.74)
  Week 36 | 2 (24.15) | 0 (15.61)
  Week 48 | 1 (24.25) | 1 (15.21)
  Week 60 | 3 (19.47) | 1 (16.37)
  Week 72 | 3 (20.22) | 1 (15.12)
  Week 84 | 2 (20.43) | 1 (17.27)
  Week 96 | 1 (25.46) | 0 (12.73)

50. Primary Outcome: Safety and Tolerability in Terms of Abnormal ECG, Abnormalities
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 24 | 0 (24.02) | 0 (15.74)
  Final Visit | 0 (25.46) | 0 (12.73)

51. Primary Outcome: Safety and Tolerability in Terms of Abnormal Physical Exams, Cardiovascular
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 1 (15.61)
  Week 48 | 0 (24.25) | 1 (15.21)
  Week 60 | 0 (19.47) | 1 (16.37)
  Week 72 | 0 (20.22) | 1 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

52. Primary Outcome: Safety and Tolerability in Terms of Abnormal Physical Exams, General Appearance
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 1 (23.57) | 2 (15.02)
  Week 6 | 1 (23.57) | 2 (15.32)
  Week 12 | 1 (23.90) | 2 (14.94)
  Week 18 | 1 (23.56) | 2 (14.83)
  Week 24 | 1 (24.02) | 2 (15.74)
  Week 36 | 1 (24.15) | 2 (15.61)
  Week 48 | 1 (24.25) | 2 (15.21)
  Week 60 | 1 (19.47) | 2 (16.37)
  Week 72 | 1 (20.22) | 2 (15.12)
  Week 84 | 1 (20.43) | 2 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

53. Primary Outcome: Safety and Tolerability in Terms of Abnormal Physical Exams, Head and Neck
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 1 (15.02)
  Week 6 | 0 (23.57) | 1 (15.32)
  Week 12 | 0 (23.90) | 1 (14.94)
  Week 18 | 0 (23.56) | 1 (14.83)
  Week 24 | 0 (24.02) | 1 (15.74)
  Week 36 | 0 (24.15) | 1 (15.61)
  Week 48 | 0 (24.25) | 1 (15.21)
  Week 60 | 0 (19.47) | 1 (16.37)
  Week 72 | 0 (20.22) | 1 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

54. Primary Outcome: Safety and Tolerability in Terms of Abnormal Physical Exams, Musculoskeletal/Extremities
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 1 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

55. Primary Outcome: Safety and Tolerability in Terms of Abnormal Physical Exams, Skin
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 3 (23.57) | 2 (15.02)
  Week 6 | 3 (23.57) | 2 (15.32)
  Week 12 | 3 (23.90) | 2 (14.94)
  Week 18 | 3 (23.56) | 2 (14.83)
  Week 24 | 3 (24.02) | 2 (15.74)
  Week 36 | 3 (24.15) | 2 (15.61)
  Week 48 | 3 (24.25) | 2 (15.21)
  Week 60 | 2 (19.47) | 2 (16.37)
  Week 72 | 2 (20.22) | 2 (15.12)
  Week 84 | 2 (20.43) | 1 (17.27)
  Week 96 | 2 (25.46) | 1 (12.73)

56. Primary Outcome: Safety and Tolerability in Terms of Abnormal Vital Signs
Time Frame: 96 weeks
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 4 | 5
participants
  Baseline | 0 (23.57) | 0 (15.02)
  Week 6 | 0 (23.57) | 0 (15.32)
  Week 12 | 0 (23.90) | 0 (14.94)
  Week 18 | 0 (23.56) | 0 (14.83)
  Week 24 | 0 (24.02) | 0 (15.74)
  Week 36 | 0 (24.15) | 0 (15.61)
  Week 48 | 0 (24.25) | 0 (15.21)
  Week 60 | 0 (19.47) | 0 (16.37)
  Week 72 | 0 (20.22) | 0 (15.12)
  Week 84 | 0 (20.43) | 0 (17.27)
  Week 96 | 0 (25.46) | 0 (12.73)

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=9)
Nasopharyngitis (Infections and infestations) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon completion of the Clinical Trial (CT), the Principal Investigator (PI) may prepare the data derived from the CT for publication or presentation. Material should be submitted to the Sponsor for review prior to review or submission for publication. Publications from individual sites must not precede the primary manuscript, but if published within twelve months after completion of the CT, the PI has the right to publish or present the methods and results of the CT.